CLINICAL TRIAL: NCT03014557
Title: China REgistry of WATCHMAN Left Atrial Appendage Closure for Non-valvular Atrial Fibrillation
Brief Title: China REgistry of WATCHMAN
Acronym: CREW
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fu Wai Hospital, Beijing, China (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Shu Zhang, Director of Department of Arrhythmia, Fu Wai Hospital, Beijing, China
Other Study IDs: T2016-ZX021
Record Dates: First submitted 2017-01-04; First posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage Closure
Keywords: atrial fibrillation; left atrial appendage closure; WATCHMAN
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- WATCHMAN: subjects with non-valvular atrial fibrillation intended to be implanted with a WATCHMAN left atrial appendage closure device
  Interventions: Device: left atrial appendage closure device implantation

INTERVENTIONS:
Device: left atrial appendage closure device implantation — to permanently implant a WATCHMAN left atrial appendage closure device through trans-catheter approach

SUMMARY:
This registry is designed to observe the safety and effectiveness of WATCHMAN left atrial appendage closure technology in a Chinese population.

DETAILED DESCRIPTION:
In this prospective, multi-center, single arm observational study, 413 patients with non-valvular atrial fibrillation intended to be implanted with a WATCHMAN device based on real clinical practice will be enrolled. Enrolled subjects will be followed up for 5 years.Primary endpoints include stroke, systematic embolism, cardiovascular death, and procedure or device related complications, etc.

ELIGIBILITY:
Inclusion Criteria:

Non-valvular atrial fibrillation patient with CHA2DS2-VASC≥2, and with any one of the following items:

1. not suitable for long-term anti-coagulation therapy;
2. stroke or embolism events in spite of warfarin treatment with intended INR
3. HAS-BLED≥3

Exclusion Criteria:

Patient with any one of the following items will be excluded from the study:

1. clinical exclusion criteria (any of the items) a congestive heart failure NYHA IV, b atrial septum defect, ASD surgery or closure c cardioversion or catheter ablation is planned within 30 days d with mechanic valve e left atrial appendage resection f heart transplantation g symptomatic jugular artery disease h previous stroke or TIA within 30 days i long term warfarin therapy is needed or contraindicated to warfarin j contraindicated to aspirin or clopidogrel k enrolled in other cardiac device or medicine trials l pregnant women or plan to pregnant during the study period m estimated life < 5 years

2 Echocardiography exclusion criteria (any of the items) a LVEF<30% b thrombus or spontaneous echo imaging detected within two days prior to procedure c patent foramen ovale d cardiac tumor e left atrial appendage orifice diameter >32mm or < 17mm f the depth of left atrial appendage is less than the width g prominent mitral stenosis (area <1.5cm2)

3 subject is not able to or will not complete the follow ups as planned

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: non-valvular atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 413 (Estimated)
Dates: Start 2016-11; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
all-cause death, ischemic stroke, systemic embolism, or device or procedure related events | between the time of enrollment and within 7 days of the procedure or by hospital discharge, whichever is later
  events requiring open cardiac surgery or major endovascular intervention such as pseudoaneurysm repair, AV fistula repair, or other major endovascular repair.
composite endpoint of hemorrhagic stroke, ischemic stroke, systemic embolism or cardiovascular/unexplained death. | 2 years

SECONDARY OUTCOMES:
Implantation success rate. | procedure
  Implantation success is defined as successful delivery and release of WATCHMAN into the LAA including successful recapture and retrieval if necessary.
Ischemic stroke or systemic embolism | excluding the first 7 days post enrollment.
All Major Complications. | up to 5 years
  Major complication is defined as death, stroke, MI or any other serious adverse events related to the device or procedure.
All-cause death. | up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No